CLINICAL TRIAL: NCT07377929
Title: Intradetrusor Onabotulinumtoxin A (Botox) at the Time of Transurethral Resection of the Prostate or Transurethral Waterjet Ablation of the Prostate for Mixed Lower Urinary Tract Symptoms
Status: Recruiting | Type: Observational
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Will Fuller, Principal Investigator, Benaroya Research Institute
Other Study IDs: IRB24-069
Record Dates: First submitted 2025-03-24; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Benign Prostatic Hypertrophy (BPH); Lower Urinary Track Symptoms
Keywords: lower urinary tract symptoms (LUTS); benign prostatic hypertrophy (BPH); overactive bladder syndrome (OAB); Transurethral resection of the prostate (TURP); Transurethral Waterjet Ablation of the Prostate (Aquablation); Botox
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Group: This group will contain men (>=18 years) and will be scheduled to undergo TURP or Aquablation and Botox procedure.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — * 1 week post-operative visit for: trial of void, to assess for rates of postoperative urinary retention.
  * 4 and 12 week post-operative visits for: post void residual assessment via bladder scan, AUA symptom score, PGI-I, UDI-6, and VM Post Procedure questionnaires will be administered
  * Hospitalization readmission rates, urinary retention episodes will also be recorded.
  Other Names: AUA symptom score; PGI-I; UDI-6; VM Post Procedure questionnaires; post void residual assessment via bladder scan

SUMMARY:
Patients with longstanding obstructive lower urinary tract symptoms (LUTS) due to benign prostatic hypertrophy (BPH) can also develop symptoms of overactive bladder syndrome (OAB). Transurethral resection of the prostate (TURP) and Transurethral Waterjet Ablation of the Prostate (Aquablation) are amongst the gold standard surgical treatments for BPH. However, in the immediate post-operative period, TURP and Aquablation can also include OAB-like symptoms, including urinary frequency and urgency. For men with baseline OAB symptoms, this initial worsening of symptoms can be distressing.

Botox is an FDA approved medication with on-label indications to treat overactive bladder.

The purpose of this study is to evaluate the outcomes of men who have Botox concurrent with their TURP or Aquablation.

ELIGIBILITY:
Inclusion Criteria:

1. Male >= 18 years of age and being scheduled to undergo TURP or Aquablation and Botox procedure.
2. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

   Exclusion Criteria:
3. Non-English speaking
4. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
5. History of receiving Botox in the bladder, within the previous 12 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be identified by patients visiting the Virginia Mason Medical Centers Urology department.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
To identify whether concurrent Botox and TURP or Aquablation are effective at reducing post-operative irritative voiding symptoms. | 4 months
  This will be measured using Postoperative Urinary Retention (POUR):
  At 1 week post-operative visit for trial of void to assess for rates of postoperative urinary retention.
  At 4 and 12 week post-operative visits for post void residual assessment

SECONDARY OUTCOMES:
To identify whether concurrent Botox and TURP or Aquablation lead to longer hospitalizations. | 4 months
  Analyzing admission data to determine if there are any changes to the hospital admission rates.
To identify whether concurrent Botox and TURP or Aquablation lead to higher rates of urinary retention. | 4 months
  Analyzing admission data to determine if there are any changes to the urinary retention episodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Mason Franciscan Health, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Virginia Mason Urology providers will identify patients for potential study participation.
  Informed consent will be obtained for all subjects who wish to participate in this trial. Upon consent, study staff will obtain baseline and demographic data, administer AUA symptom score and the UDI-6. At follow up visits, the AUA symptom score, UDI-6, PGI-I, and VM post-procedure questionnaire will be obtained for participating patients. Additional data points under study will be obtained from the subject's electronic medical record.
  All study data will be entered into a secure password-protected clinical research database maintained on a Virginia Mason computer. No PHI will be transferred outside of Virginia Mason.

REFERENCES:
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Yap TL, Cromwell DA, Brown C, van der Meulen J, Emberton M. The relationship between objective frequency-volume chart data and the I-PSS in men with lower urinary tract symptoms. Eur Urol. 2007 Sep;52(3):811-8. doi: 10.1016/j.eururo.2007.01.013. Epub 2007 Jan 12. PMID 17276583
- [Background] Palnaes H.C., Klarskov P.: The accuracy of the frequency-volume chart: comparison of self-reported and measured volumes. Br J Urol 1998; 81: pp. 709-711
- [Background] Zillioux J, Welk B, Suskind AM, Gormley EA, Goldman HB. SUFU white paper on overactive bladder anticholinergic medications and dementia risk. Neurourol Urodyn. 2022 Nov;41(8):1928-1933. doi: 10.1002/nau.25037. Epub 2022 Sep 6. PMID 36066046
- [Background] Al-Shaiji TF. Intradetrusor injection of botulinum toxin for the management of refractory overactive bladder syndrome: an update. Surg Innov. 2013 Aug;20(4):351-5. doi: 10.1177/1553350612460125. Epub 2012 Sep 10. PMID 22964263
- [Background] Gormley EA, Lightner DJ, Burgio KL et al: Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline. J Urol 2012; 188: 2455
- [Background] Lightner DJ, Gomelsky A, Souter L et al: Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU Guideline amendment 2019. J Urol 2019; 202: 558
- [Background] Kim SJ, Al Hussein Alawamlh O, Chughtai B, Lee RK. Lower Urinary Tract Symptoms Following Transurethral Resection of Prostate. Curr Urol Rep. 2018 Aug 20;19(10):85. doi: 10.1007/s11934-018-0838-4. PMID 30128964
- [Background] Cornu JN, Grise P. Is benign prostatic obstruction surgery indicated for improving overactive bladder symptoms in men with lower urinary tract symptoms? Curr Opin Urol. 2016 Jan;26(1):17-21. doi: 10.1097/MOU.0000000000000249. PMID 26574877
- [Background] Gilling PJ, Barber N, Bidair M et al. Five-year outcomes for Aquablation therapy compared to TURP: results from a double-blind, randomized trial in men with LUTS due to BPH. Can J Urol. 2022 Feb;29(1):10960-10968
- [Background] Lerner LB, McVary, KT, Barry MJ et al: Management of lower urinary tract symptoms attributed to benign prostatic hyperplasia: AUA Guideline part II, surgical evaluation and treatment . J Urol 2021; 206: 818
- [Background] Lerner LB, McVary, KT, Barry MJ et al: Management of lower urinary tract symptoms attributed to benign prostatic hyperplasia: Make it since she anything that change in point being between resident it level at and exchanged between if something to do it and it would not is I am still and she feels with the numbers she old Knee she I put there is no Guideline part I, initial work-up and medical management. J Urol 2021; 206: 806.
- [Background] Chen LC, Kuo HC. Pathophysiology of refractory overactive bladder. Low Urin Tract Symptoms. 2019 Sep;11(4):177-181. doi: 10.1111/luts.12262. Epub 2019 Mar 22. PMID 30900373
- [Background] Ng M, Leslie SW, Baradhi KM. Benign Prostatic Hyperplasia. 2024 Oct 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK558920/ PMID 32644346

DOCUMENTS (2):
  • Study Protocol (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT07377929/Prot_000.pdf
  • Informed Consent Form (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT07377929/ICF_001.pdf